CLINICAL TRIAL: NCT03778996
Title: Phase 2 Clinical Trial to Evaluate Efficacy and Safety of SM-88 Used With Methoxsalen, Phenytoin, and Sirolimus (MPS) as Maintenance Therapy Following Standard Treatments for Ewing's Sarcoma or as Salvage Therapy for Advanced Sarcomas
Brief Title: SM-88 Maintenance Therapy for Advanced Ewing's Sarcoma and as Salvage Therapy for Sarcoma
Acronym: HopES
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Oncology Research Center, LLC (Other)
Collaborators: Tyme, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SM-88-JAF-16
Record Dates: First submitted 2018-12-06; First posted 2018-12-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma, Ewing; Sarcoma
Keywords: Ewing's Sarcoma; Locally advanced sarcoma; Metastatic sarcoma; SM-88; D.L-alpha-metyrosine
MeSH Terms: conditions — Sarcoma, Ewing; Sarcoma | interventions — Methoxsalen; Phenytoin; Sirolimus; racemetyrosine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maintenance Treatment: Ewing's Sarcoma (Experimental): Combination metyrosine-derivative, low-dose methoxsalen, phenytoin and sirolimus
  Interventions: Drug: Combination metyrosine-derivative, low-dose methoxsalen, phenytoin and sirolimus (MPS)
- Salvage Treatment: Sarcoma (Experimental): Combination metyrosine-derivative, low-dose methoxasalen, phenytoin and sirolimus
  Interventions: Drug: Combination metyrosine-derivative, low-dose methoxsalen, phenytoin and sirolimus (MPS)

INTERVENTIONS:
Drug: Combination metyrosine-derivative, low-dose methoxsalen, phenytoin and sirolimus (MPS) — Daily oral combination therapy for cancer
  Other Names: SM-88

SUMMARY:
The primary objective is to evaluate the efficacy of SM-88, a combination metabolic cancer treatment, in two study cohorts:

* Clinically advanced Ewing's Sarcoma patients who have not progressed at the conclusion of systemic treatment
* Clinically advanced sarcoma patients in the salvage treatment setting

Up to 24 efficacy evaluable patients (up to 12 per cohort) will be enrolled. Study patients will receive oral SM-88, with scheduled safety and efficacy evaluations.

DETAILED DESCRIPTION:
This prospective, open-label, two stage, pilot phase 2 trial evaluates the efficacy and safety of SM-88 in two cohorts of patients: 1) as maintenance therapy following standard primary or palliative treatments for Ewing's sarcoma patients with high risk of relapse or disease progression; and 2) as salvage therapy for patients with clinically advanced sarcomas.

The primary objective is to evaluate the efficacy of SM-88, a combination metabolic cancer treatment, measured as positive efficacy events, including overall response, maintaining stable disease for ≥ 3 months, or progression free survival at least 1.5 times longer than the last prior line of treatment.

Eligible patients will receive daily oral treatment with SM-88, which consists of D,L-alpha-metyrosine, used with methoxsalen, phenytoin, and sirolimus in continuous treatment cycles of 28 days. Treatment will continue until: 1) Symptomatic, clinical progression with radiographic progressive disease; 2) 48 weeks after documented complete response; or 3) evidence of unacceptable toxicity, or other decision to discontinue treatment

ELIGIBILITY:
Key Inclusion Criteria:

1. Ability to understand and willingness to provide written informed consent to participate in this study
2. ≥12 years of age
3. Diagnosis:

   1. Maintenance treatment cohort: Histologic or cytologic diagnosis of Ewing's sarcoma, including non-resected, locally advanced or metastatic disease
   2. Salvage treatment cohort: Non-resected, locally advanced or metastatic sarcoma (including Ewing's sarcoma) for which there is no standard of care treatment and no curative other option
4. Radiographic disease assessment within 35 days prior to enrollment and planned treatment start with study drug
5. Prior treatment:

   1. Maintenance treatment cohort : 1-3 prior lines of systemic treatment (including current treatment)
   2. Salvage cohort: Any number of prior treatments
6. Maintenance treatment cohort only: Patient completed current line of treatment (systemic, surgery, radiation) prior to enrollment, without disease progression as compared to baseline AND has achieved at least one of the following

   1. CR in response to current second or third line treatment
   2. PR in response to current line of treatment (after at least 4 cycles, if treatment included systemic therapy)
   3. SD in response to current line of treatment (after at least 4 cycles, if treatment included systemic therapy)
7. Measurable disease, except for patients in Cohort A who have achieved CR at the conclusion of current 2nd or 3rd line of treatment
8. ECOG performance status 0-2
9. Adequate organ function defined as all laboratory parameters ≤ Grade 2 NCI CTCAE criteria
10. Patients must be able to swallow and retain whole capsules

Key Exclusion Criteria:

1. Systemic anticancer agents within 14 days prior to treatment on study
2. Major surgery within 30 days
3. Prior treatment with SM-88
4. Any screening laboratory, electrocardiogram (ECG), other clinical finding, comorbidity or clinical history that, in the opinion of the investigator, indicates an unacceptable risk for patient to participate in the study or would limit patient's ability to comply with study requirements
5. History of any drug allergies or significant adverse reactions to any of the components of SM-88
6. History of light sensitive diseases for which methoxsalen would be contraindicated
7. Current or anticipated treatment with a contraindicated medication
8. Evidence of viral infections including human immunodeficiency virus (HIV), hepatitis B, and hepatitis C

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2027-12-19 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Every 3 months for up to 2 years
  Complete response (CR) + partial response (PR) as evaluated using RECIST 1.1
Stable Disease for at Least 3 Months | Every 3 months for up to 2 years
  Stable disease (SD) as evaluated using RECIST 1.1
Progression Free Survival on Study of at Least 1.5 Times the Duration of PFS for the Last Prior Treatment | Every 3 months for up to 2 years
  From date of enrollment until the date of first documented progression, as evaluated using RECIST 1.1, or date of death, whichever occurs first

SECONDARY OUTCOMES:
Duration of Response | Every 3 months for up to 2 years
  From date of CR or PR until the date of first documented progression, as evaluated using RECIST 1.1
Overall Survival | Every 3 months for up to 2 years
  From date enrollment until the date of death
Clinical Benefit Rate | Every 3 months for up to 2 years
  CR+PR+SD as evaluated using RECIST 1.1
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5 | From date of enrollment until 28 days after last treatment with SM-88
  Adverse events will be assessed at each visit and at unscheduled visits as clinically indicated

CONTACTS AND LOCATIONS:
Overall Officials: Sant P Chawla, MD, Principal Investigator — Sarcoma Oncology Research Center
Locations (1):
- Sarcoma Oncology Research Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sarcoma Oncology Research Center — https://sarcomaoncology.com/